CLINICAL TRIAL: NCT05635097
Title: Remote Weight Management Program for Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00002292
Record Dates: First submitted 2022-11-10; First posted 2022-12-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group intervention (Other): One group without comparator
  Interventions: Behavioral: Motivational Interviewing counseling on the Mediterranean diet and weight checks at regular intervals

INTERVENTIONS:
Behavioral: Motivational Interviewing counseling on the Mediterranean diet and weight checks at regular intervals — Each participant will meet virtually on Zoom with the DNP project leader and receive 1:1 counseling on pairing the Repnho smart scale and tape measure with the Renpho application. The expectations of the weight management program will be explained in detail during the first session, which will last one hour (session one= week zero). The weight loss goal will be at least 1-2 pounds per week as recommended by the Centers for Disease Control and Prevention (CDC) (2022).

SUMMARY:
The purpose of the research project is to see if counseling on the Mediterranean diet combined with motivational interviewing via a telemedicine platform (Zoom) while using smart technology ("smart" scales and tape) improves participants' weight loss, reduces waist circumference, and improves satisfaction with their care.

DETAILED DESCRIPTION:
The investigators will evaluate a formal remote weight management and follow-up program, utilizing a technology-based intervention using the Renpho application paired with a smart scale and smart tape measure. The primary communication technologies will be the REDCap and Zoom platforms.

Renpho's smart body fat scale and tape measure are health applications that sync with fitness applications such as Apple Health, MyFitnessPal, Fitbit, and Samsung Health. The Renpho Bluetooth-enabled smart scale and smart tape devices will allow participants to sync with the Renpho application on their smartphone to automatically upload data such as weight, BMI, and WC to their phone. The project leader will review participants' self-reported weights and WC fortnightly. The participants will be asked to complete a post-participation satisfaction survey that includes a 5-point scale ("strongly agree", "agree", "neutral", "disagree:", to "strongly disagree") Likert-style questions.

Expected Outcomes. The primary outcomes for this eight-week intervention are to achieve a clinically significant reduction in weight of at least 5-10 % and at least 2.5 inches reduction in WC per participant from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a clinical diagnosis of obesity (BMI ≥30 kg/m2),
2. Age of 18 years or older,
3. English-speaking participants with access to a smartphone device
4. At least one cardiovascular risk factor (at least one clinical diagnosis of the following conditions: hypertension, dyslipidemia, type 2 diabetes, pre-diabetes, sleep apnea, family history of heart disease, cigarette smoking, inactivity, preeclampsia, gestational diabetes, gestational hypertension, preterm birth, rheumatological diseases, or premature menopause).

Exclusion Criteria:

1. Must not be taking medications specifically for weight loss or currently participating in a weight loss program,
2. Must not be pregnant or breast-feeding,
3. Women without a clinical diagnosis of obesity (BMI < 30 kg/m2)
4. Must not have lost >3 kg body weight or dramatically changed physical activity patterns within the past six months,
5. Clinical diagnosis of eating disorders
6. Clinical diagnosis of uncontrolled hypertension or neurological or psychological disorders
7. Must not have any obesity-related surgery within the past six months (i.e., gastric bypass).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Enrollment: 30 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Weight change (in pounds) | 8 weeks
  Weight of at least 5-10 % per participant from baseline

SECONDARY OUTCOMES:
Waist circumference change (in inches) | 8 weeks
  At least 2.5 inches change per participant from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Depends on positive/negative results